CLINICAL TRIAL: NCT01962129
Title: Clinical and Molecular Characterisation of Orofaciodigital Syndromes and Other Clinical Phenotypes Secondary to Mutations in the OFD1 Gene
Acronym: OFD1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Thauvin PHRC N 2010
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Orofaciodigital Syndromes
MeSH Terms: conditions — Orofaciodigital Syndromes

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients affected by a syndrome OFD
  Interventions: Biological: Sampling of blood
- Patients AFFECTED BY A SEVERE MENTAL RETARDATION SYNDROMIQUE
  Interventions: Biological: Sampling of blood

INTERVENTIONS:
Biological: Sampling of blood

SUMMARY:
The aim of this multicentre study will be to better describe the clinical characteristics and the etiological bases of patients with OFD syndrome by identifying new genes involved in OFD syndrome. These results will make it possible, from patients who have been clearly identified from a clinical, cytogenetic and molecular point of view, to determine a study strategy in such patients. The data obtained will be used to guide clinical geneticists in genetic counselling for patients and their families.

Identification of the molecular bases of the different OFD syndromes will make it possible to determine whether or not they belong to the group of ciliopathies like type I OFD and to understand their physiopathological bases.

This study will also make it possible to better characterise the phenotype of boys with syndromic mental retardation related to the OFD1 gene and thus to define the clinical criteria of the study of this gene in boys with mental retardation.

The complete absence of knowledge concerning the genetic bases of OFD syndromes, apart from type I, the presence of a large collection of samples from patients with OFD syndrome at Dijon CHU, the recognition of the diagnostic laboratory for syndromic OFD at the international level as well as the technical platform and expertise in molecular cytogenetic methods including CGH-array and molecular genetics (sequencing, quantitative PCR, fragment analysis) at the Cytogenetics and Molecular Biology laboratories at Dijon CHU justify the implementation of such a study in 2010.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Study the molecular bases of OFD syndromes Patients from whom samples have been collected - declaration to the Ministry in progress Patients with an OFD syndrome with samples in the collection DC-2009-1045 and for which the declaration to the Ministry is in progress, will be included in this study. Indeed, the blood samples of 65 patients have been sent to us since 2002 for the study of the OFD l gene thanks to national and international recruitment: 35 presented clinical signs more or less associated with a mode of transmission suggesting OFD l syndrome and 30 presented other forms of OFD (OFDII, OFDVI, OFDVII, OFDVIII and OFDIX) or a polymalformative syndrome with OFD involvement (OFD+). We therefore constituted a second collection of DNA samples from 33 patients with OFD syndrome or a polymalformative syndrome with OFD involvement, who presented neither a mutation nor a rearrangement of the OFD1 gene.

The clinical data are already available from Doctor Christel Thauvin-Robinet, who is responsible for this collection. These patients have signed a non-opposition form allowing the use of their blood samples for research on OFD syndromes. These patients will therefore be included in this new study without the need for new consent. Only an information letter will be sent to them (annexe 4A)

Newly-included patients The inclusion criteria for patients are principally clinical and/or paraclinical, based on the clinical investigation usually conducted in the follow-up of these patients. Every index case must present an OFD syndrome with normal results for the study of the OFD1 gene by direct sequencing of genomic DNA and a search for major rearrangements using quantitative PCR. The index cases could be children (from birth onwards) or adults, male or female with sporadic or familial syndromes.

Patients will be recruited by the clinical investigators of this study. These patients could be:

* patients already known by the investigator, who will contact the patient to invite them to take part in the research,
* or new patients seen during a consultation in the first year of the study (inclusion period) The clinical dossier that accompanies each sample will include a case report form, a family tree, photographs of the patient a signed written informed consent form Symptomatic and asymptomatic relatives may also be included in our study, once their written informed consent has been provided, so as to exclude polymorphism using CGH-array or molecular biology, or to confirm the segregation of a mutation.

Minors will only be included in our study if they are symptomatic. All of those who take part in this research, whether they are patients or healthy or asymptomatic relatives have to be covered by a national health insurance agency.

Group 2: Study of the form of syndromic X-linked mental retardation secondary to mutations in the OFD1 gene Preexisting patient cohorts

Two different types of populations could be included:

* Boys with Joubert syndrome with cerebellar hypoplasia at the origin of the "molar tooth" sign on cerebral MRI and a negative result for mutations in the genes involved in Joubert syndrome as described by Doctor Burglen (Hospital Trousseau, APHP)
* Boys with a phenotype that could be linked to mutations in the OFD1 gene:

  * A cohort of boys with polydactyly+/- juvenile retinitis pigmentosa or obesity who were screened negative for BBS gene mutations recruited through Professor Dollfus (CHU Strasbourg)
  * A cohort of males with severe macrocephaly (>+4SD) with negative screening for mutations in the GPC3 gene recruited through Doctor Rossignol (CHU Trousseau, Paris) and Doctor Raynaud (CHU Tours).
  * A cohort of males with recurrent pulmonary infections, macrocephaly (>+4SD) and negative screening for mutations in the MECP2 gene recruited through Doctor Philippe (CHU Nancy), Doctor Badens (CHU Marseille), Professor Bieth (CHU Toulouse) and Professor Touraine (CHU St Etienne).

The clinical dossier that accompanies each DNA sample will include a case report form, a family tree, photographs of the patient a signed written informed consent form

Newly-included patients The inclusion criteria for patients are principally clinical and/or paraclinical, based on the clinical investigation usually conducted in the follow-up of these patients. All of the index cases will be males who must present: (1) Joubert syndrome with normal results for the genes responsible for Joubert syndrome or (3) syndromic mental retardation more or less associated with polydactyly, obesity, macrocephaly, pigmentary retinopathy, recurrent infections and/or the "molar tooth" sign on cerebral MRI. Index cases could be infants (from birth onwards) or adults, sporadic or familial cases with a mode of transmission compatible with X-linked inheritance.

Patients will be recruited by the clinical investigators of this study. These patients could be:

* patients already known by the investigator, who will contact the patient to invite them to take part in the research,
* or new patients seen during a consultation in the first year of the study (inclusion period) The clinical dossier that accompanies each sample will include a case report form, a family tree, photographs of the patient a signed written informed consent form Symptomatic and asymptomatic relatives may also be included in our study, once their written informed consent has been provided, so as to exclude polymorphism using CGH-array or molecular biology, or to confirm the segregation of a mutation.

Minors will only be included in our study if they are symptomatic. All of those who take part in this research, whether they are patients or healthy or asymptomatic relatives have to be covered by a national health insurance agency.

Exclusion criteria:

Patients will be excluded from the study if the clinical data do not meet the criteria defined above.

Patients with OFD syndrome in whom sequencing of the exons or exon-intron junctions of the OFD1 gene of genomic DNA and the search for major rearrangements quantitative PCR identify a causal mutation will not be included in this study.

The following patients will also be excluded from the study:

* those who do not wish to provide a blood sample,
* those who have not provided written informed consent,
* those without national health insurance,
* those in custody following a legal or administrative decision.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orofaciodigital Syndromes type I, type VII or other orofaciodigital syndromes
Sampling Method: Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Blood Samples | baselines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France